CLINICAL TRIAL: NCT06758570
Title: The Modulatory Effects of Dietary Fibres on the Composition and Function of the Gut Microbiome- A Dose-response Study
Brief Title: Effect Dietary Fibre Supplementation on Gut Microbiota Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Simpson (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Organization: University of Nottingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FMHS 302-0621(Dose response)
Record Dates: First submitted 2024-08-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Diet, Healthy; Systemic Inflammatory Response
Keywords: Dietary intervention; Gut microbiome; Dose- response; Systemic inflammation

STUDY DESIGN:
Intervention Model Description: Dose-response study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose response effect of Pectin (Experimental): In order to investigate the dose-response effect of dietary pectin fibre, pectin was provided to healthy volunteers in increasing doses of 5g, 10g and 15g for a period of 2 weeks each with samples and data collected prior to each dosing period.
  Interventions: Dietary Supplement: Pectin dosages

INTERVENTIONS:
Dietary Supplement: Pectin dosages — 15 individuals were provided with increasing doses of pectin: 5g for 2 weeks 10g for 2 weeks 15 for 2 weeks

SUMMARY:
The study involves taking pectin fibre at increasing doses ranging from 5g, 10g and 15g for a total period of 6 weeks with the increase every 2 weeks. Study subjects will be healthy volunteers recruited from the University and local population and will be asked to attend the laboratory on 4 occasions; at the start of the intervention and every 2 weeks, at the end of each dosing period. At each study visit (~3hrs), participants will be asked to provide a stool and blood sample and will have blood pressure measured. In the week before each study visit, participants will record their food intake.

DETAILED DESCRIPTION:
The study aims to assess the optimal dosage of pectin required to see beneficial effects on inflammation and gut microbiome composition. 15 healthy, non-obese volunteers will be recruited following a successful medical screening. Between recruitment and first study visit, and at the end of each dosing period (before each study visit), participants will be asked to complete a dietary record (4 days), to collect a stool sample on the day before the study visit and to fast from midnight the night before this visit.

At both study visits, participants will have weight, hip/waist circumference and blood pressure measured. They will be asked to complete some questionnaires. After completion of the first study day, participants will be provided with the required dosage of pectin for the 2-week dosing period. They will be given the required doses of pectin portioned in individual sachets, with instructions to add the contents of one sachet a day to juice, smoothies or water and to consume immediately. Study visits will be scheduled at the end of every 2-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participant eligibility includes those aged >18 years who have a body mass index (BMI) between 18.5 and 39.9 kg/m2

Exclusion Criteria:

* Have psychosocial or gastrointestinal (e.g. malabsorptive conditions such as IBS/IBD, coeliac)
* Are taking the following medications: immunosuppressants, anti-histamines, amiodarone and/or perhexiline
* Are currently following or anticipated to commence a specialised commercially available weight loss diet and/or program/ taking prebiotic supplements
* Pregnant or breast feeding
* History or current psychiatric illness
* History or current neurological condition (e.g. epilepsy)
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in microbiome profile | 6 weeks
  Change in microbiome profile, assessed using 16s RNA sequencing analysis of faecal samples provided at the start (pre-intervention) and end of every dosing period (i.e. 2 weeks)
Change in inflammatory profile | 6 weeks
  Change in circulating markers of inflammation measured by ELISAs in serum samples collected at the start (pre-intervention) and end of every dosing period (i.e. 2 weeks).
Changes in short chain fatty acids (SCFAs) | 6 weeks
  Change in serum SCFAs measured by mass spectrometry at the start (pre-intervention) and end of every dosing period (i.e. 2 weeks).

SECONDARY OUTCOMES:
Change in systolic blood pressure (lying to standing) pre intervention | 6 weeks
  Change in systolic blood pressure (measured after 3 minutes of lying down and after 1 minute of standing), at pre-intervention study visit.
Dose response change in Short Form Health Survey (SF36) Questionnaire aggregated normalised 'physical' score | 6 weeks
  Change in 'SF36' Questionnaire aggregated 'physical' score (normalised to UK population) calculated according to standard procedures (min 0, max 100), with higher score indicating better physical wellbeing; measured at the start and the end of each dosing period
Dose response change in Short Form Health Survey (SF36) Questionnaire aggregated normalised 'mental' score | 6 weeks
  Change in 'SF36' Questionnaire aggregated 'mental' score (normalised to UK population) calculated according to standard procedures (min 0, max 100), with higher score indicating better physical wellbeing; measured at the start and the end of each dosing period
Dose response change in Pittsburgh Sleep Quality Index (PSQI) | 6 weeks
  Change in PSQI score (min score 0, max 21), measured at the start and the end of each dosing period, with higher score indicating poorer sleep quality
Dose response change in Hospital Anxiety and Depression scores (HADS) | 6 weeks
  Change in anxiety score (min 0, max 3 which higher scores indicating higher anxiety like symptoms) and depression scores (min 3, max 0 which lower scores indicating higher depressive like symptoms), measured at the start and at the end of each dosing period
Change in systolic blood pressure (lying to standing) post every dosing period | 6 weeks
  Change in systolic blood pressure (measured after 3 minutes of lying down and after 1 minute of standing), at the end of each dosing period (every 2 weeks)
Change in diastolic blood pressure (lying to standing) post every dosing period | 6 weeks
  Change in diastolic blood pressure (measured after 3 minutes of lying down and after 1 minute of standing), at the end of each dosing period (every 2 weeks)
Change in diastolic blood pressure (lying to standing) at pre intervention study visit | 6 weeks
  Change in diastolic blood pressure (measured after 3 minutes of lying down and after 1 minute of standing), pre intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ana Valdes, Professor, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom